CLINICAL TRIAL: NCT04702477
Title: An Innovative Approach With Group Counseling and Mindfulness Training Among Prediabetes Patients
Brief Title: Mindfulness Training and Group Counseling Among Prediabetes and Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clemson University (Other)
Collaborators: University of California, Los Angeles (Other); Prisma Health-Upstate (Other)
Responsible Party: Principal Investigator, Heidi Zinzow, Professor of Psychology, Clemson University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00076863
Record Dates: First submitted 2020-11-23; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-12

CONDITIONS: Stress; Diabetes; Pre-Diabetes; Health Behavior; Quality of Life
Keywords: Stress; Mindfulness; Diabetes; Pre-Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance; Health Behavior | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: This is a single-arm, paired-sample pilot intervention study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Only Arm (Experimental): This is a single-arm, paired-sample pilot intervention study among participants with pre-diabetes or diabetes. Goal to integrate a MBSR intervention into a group-based, lifestyle intervention among patients with prediabetes or diabetes in the primary care setting
  Interventions: Behavioral: Mindfulness Based Stress Reduction

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — Mindfulness Based Stress Reduction (MBSR) is a well-documented approach to reduce participants' stress level [19], with the existing group-based peer support, self-empowerment, and lifestyle counseling intervention. MBSR is a type of meditation therapy with the goal of actively cultivating conscious attention and awareness to enhance health benefits. This included 10 hours of intervention with groups of 3-5 people.

SUMMARY:
Examining a number of health outcomes in those with diabetes and prediabetes before and after a group-based mindfulness intervention.

DETAILED DESCRIPTION:
This is a pilot study to examine the feasibility of integrating a mindfulness-based stress reduction (MBSR) intervention in addition to an existing group-based, peer supported clinical care model (JUMP) among patients with pre-diabetes or diabetes using a mixed-method design.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English speaking
* Having a diagnosis of diabetes or prediabetes
* Participation in a previous group-based clinical care model-JUMP (as in "JUMPing into Diabetes Control")

Exclusion Criteria:

* Under 18 years old
* Non-English Speaking
* not having a diagnosis of diabetes or prediabetes
* No participation in JUMP model

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Intervention Attendance | 8-weeks while completing the intervention
  How many hours of intervention sessions an individual attended

SECONDARY OUTCOMES:
Perceived Stress Scale | Up to 3 months before intervention, immediately following intervention, one month after intervention
  Change in perceived stress measured by 4 Items to assess perceived stress where higher levels indicating higher levels of stress with a range of 4 to 20.
Depression | Up to 3 months before intervention, immediately following intervention, one month after intervention
  Change in depression scores from the Center for Epidemiologic Studies Depression Scale (CES-D), where higher scores indicate higher levels of depression with a range of 0 to 80.
Anxiety | Up to 3 months before intervention, immediately following intervention, one month after intervention
  Change in anxiety assessed using the Generalized anxiety disorder 7-item scale (GAD-7).
Medication Adherence | Up to 3 months before intervention, immediately following intervention, one month after intervention
  Change in medication adherence assessed using the 8-item Morisky Medication Adherence Scale. A higher score indicates higher adherence with a range of 0 to 8.
Perceived Health Status | Up to 3 months before intervention, immediately following intervention, one month after intervention
  Change in perceived health status assessed using a question asking participants to rate their health status on a 5-points rating scale where lower ratings indicate higher levels of perceived health status and higher ratings indicate lower levels of perceived health status.
Sleep Quality | Up to 3 months before intervention, immediately following intervention, one month after intervention
  Change in sleep quality assessed using the Pittsburgh Sleep Quality Index (PSQI) ranges from 7 to 28, with higher scores indicating worse sleep quality.
Physical Activity | Up to 3 months before intervention, immediately following intervention, one month after intervention
  Change in physical activity assessed using the Rapid Assessment of Physical Activity Scale (RAPA).
Mindfulness | Up to 3 months before intervention, immediately following intervention, one month after intervention
  Change in Mindfulness assessed using a 15-item Five-Facet Mindfulness Questionnaire (FFMQ).
HbA1C levels | Up to 3 months before intervention, immediately following intervention, one month after intervention
  HbA1C blood levels
Program satisfaction and barriers for attending sessions | Immediately following intervention
  Open ended questions to address engagement in the intervention, perceived usefulness of the MBSR, recommendations for intervention modification, what participants enjoyed most/least about the intervention, and reasons for missing intervention sessions. This is a qualitative measure, not numeric values were assigned. Based on Zgierska A, Rabago D, Zuelsdorff M, Coe C, Miller M, Fleming M. Mindfulness meditation for alcohol relapse prevention: a feasibility pilot study. J Addict Med. 2008 Sep;2(3):165-73. doi: 10.1097/ADM.0b013e31816f8546.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Shi, PhD, Principal Investigator — Clemson University
Locations (1):
- Prisma Health, Greenville, South Carolina, United States